CLINICAL TRIAL: NCT06878846
Title: The Relationship of Critical Shoulder Angle With Proprioception and Disability in Patients With Subacromial Impingement
Brief Title: The Relationship of Critical Shoulder Angle With Proprioception and Disability
Status: Completed | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Seda BAKTIR, Assist. Prof, Lokman Hekim University
Other Study IDs: LHU-FTR-ZSBD-03
Record Dates: First submitted 2025-02-28; First posted 2025-03-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Impingement Syndrome; Shoulder Impingement Syndrome; Subacromial Impingement Syndrome
Keywords: shoulder joint; critical shoulder angle; proprioception; disability
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subacromial Impingement Syndrome
  Interventions: Other: Correlation Study

INTERVENTIONS:
Other: Correlation Study — Assessment of correlation
  Other Names: Evaluation of Critical Shoulder Angle; Evaluation of Shoulder Proprioception; Evaluation of Shoulder Disability

SUMMARY:
With this study it will determined that the effect of critical shoulder angle which will be obtained from the MRI images of patients with Subacromial Impingement Syndrome on proprioception and disability level.

DETAILED DESCRIPTION:
Critical shoulder angle (CSA) is defined as the intersection angle between two lines which are drawn from inferior border of glenoid cavity to superior border of glenoid cavity and from inferior border of glenoid cavity to inferolateral border of acromion. Higher CSA is accepted a predisposing factor for degenerative shoulder diseases. Increase in CSA means more shear forces reflects on shoulder joint which also causes overload on the RC tendon. Increase of degeneration in shoulder joint may cause decreased proprioception. As a result of degeneration, the level of disability will be increased. At the end of this study, the relationship among critical shoulder angle, proprioception and disability could be more clearly interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Being between 25-70 years of age,
* Diagnosis of SIS based on physical examination (at least three positive results from the Neer, Jobe, Hawkins/Kennedy Impingement, and/or Painful Arc tests),
* Being Level I-II Subacromial Impingement (radiologic examination (MRI)),
* having painful arc between 60° and 120° during active shoulder elevation
* Having shoulder pain for 3 months.

Exclusion Criteria:

* Having a shoulder operation before.
* Having Cardiovascular, Rheumatological or Neurological Disease
* Having Cervical Spine Disease
* Having Physiotherapy Treatment in last 6 months.
* Having a trauma, fracture, total Rotator Cuff rupture, Frozen Shoulder on shoulder joint

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents with Level I-II Subacromial Impingement Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Critical Shoulder Angle | Baseline (The evaluation will be conducted only once)
  Critical Shoulder Angle is the intersection angle between two lines which are drawn from inferior border of glenoid cavity to superior border of glenoid cavity and from inferior border of glenoid cavity to inferolateral border of acromion. That will be measured from the MRI images of patients.

SECONDARY OUTCOMES:
Shoulder Proprioception | Baseline (The evaluation will be conducted only once)
  Shoulder proprioception will be evaluated 60° ve 90° ve 120° degrees of shoulder joint active-active, active-passive and passive-active manner.
  The Shoulder proprioception will be assessed using a bubble inclinometer.
Disability | Baseline (The evaluation will be conducted only once)
  The disability will be assessed by using SPADI (Shoulder Pain and disability Index). First part includes 5 questions inquiring pain status. Second part includes 8 questions inquiring activity participation status. Total score ranges between 0-100. Increase of scores reflects higher disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We are planning not to share this data not to declare the data of our participants with any third group.